CLINICAL TRIAL: NCT04671199
Title: Data Collection for Improvement of Domestic Patient Monitor
Brief Title: Collection of Anonymized Data for Improvement of Domestic Patient Monitor System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: 20111521176
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MP 3000 monitor — Additional monitoring

SUMMARY:
Collection of anonymized data for improvement of domestic patient monitor system comparison of commercial patient monitor

DETAILED DESCRIPTION:
the data from the patient will be collected as the baseline data for improvement of the domestic patient monitor system

ELIGIBILITY:
Inclusion Criteria:

* surgical patients

Exclusion Criteria:

* problem to monitor

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-25 (Estimated); Primary Completion 2021-12-24 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
anoymized data collection | during surgery
  agreement of ECG data from the 2 different patient monitor

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongnogu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided